CLINICAL TRIAL: NCT02494648
Title: Effects of Inspiratory Muscles Strengthening Among Coronary Patients on the Sleep Apnea Obstructive Syndrome (SAOS)
Brief Title: Effects of Inspiratory Muscles Strengthening Among Coronary Patients on the Sleep Apnea Obstructive Syndrome
Acronym: RICAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408189; 2015-A00030-49 (Other: ANSM)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea, Obstructive; Acute Coronary Syndrome
Keywords: Obstructive sleep apnea; Resistive inspiratory muscle training; Coronary artery disease; Cardiac rehabilitation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscles strengthening (Experimental): The device used is : POWERbreathe Fitness Plus, (POWERbreathe International Ltd, UK).
  Class I, CE labelled. POWERbreathe fitness Plus uses the technique of training against resistance to increase the strength, the power and the endurance of the respiratory muscles (diaphragm and rib cage).
  Interventions: Device: POWERbreathe Fitness Plus, (POWERbreathe International Ltd, UK) [Inspiratory muscles strengthening]
- Control (Placebo Comparator): No intervention
  Interventions: Other: Control

INTERVENTIONS:
Device: POWERbreathe Fitness Plus, (POWERbreathe International Ltd, UK) [Inspiratory muscles strengthening] — CAD patients participated in a 6-week (20 sessions of training) resistive inspiratory muscle training (RIMT) program for 10 minutes twice daily at a training intensity of 70% of maximum inspiratory pressure (MIP).
  Arms: Inspiratory muscles strengthening
Other: Control
  Arms: Control

SUMMARY:
Obstructive sleep apnea (OSA) syndrome affects up to 5% of the general population. The prevalence is multiplied by 13 in coronary artery disease (CAD) patients. Many studies have shown that OSA syndrome was the main risk factor for cardiovascular morbidity and mortality (RR = 9.1 [95%, 2.6 to 31.2]).

If the value of treatment with Continuous Positive Airway Pressure (CPAP) in symptomatic CAD patients (daytime sleepiness and/or 2 clinical symptoms with Apnea Hypopnea Index (AHI) ≥ 20) appears to be established, treatment with CPAP in asymptomatic CAD patients (with AHI> 30) may be too demanding. Alternative treatments are rare and results are highly variable. Therefore, it would be interesting to suggest other treatment modalities with moderate coronary and/or minimally symptomatic OSA syndrome.

DETAILED DESCRIPTION:
This study aims to assess the relevance of inspiratory muscles strengthening on reducing AHI in CAD patients with moderate OSA (AHI between 15 and 30).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate OSA (15 <AHI <30)
* Period between acute coronary syndrome and inclusion <60 days
* Patients included in cardiac rehabilitation

Exclusion Criteria:

* Obstructive lung disease with Tiffeneau index less than 70%.
* Restrictive lung disease with a reduction of total lung capacity (TLC)
* Treatment for OSA or clinical context (comorbidity) justifying CPAP
* Congestive heart failure, thoracic surgery by sternotomy
* Spontaneous pneumothorax
* Severe Asthma
* Ruptured eardrum, or another disease of the middle ear, or acute sinusitis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
AHI Variation | At 6 weeks
  It is the difference between the AHI at the inclusion et the AHI at 6 weeks

SECONDARY OUTCOMES:
Circumference of the neck in centimetre | At 6 weeks
  in centimetre
Epworth questionnaire to evaluate the deficit of sleep | at 6 weeks
  This questionnaire evaluates the deficit of sleep
Pittsburgh questionnaire to evaluate the quality of sleep | At 6 weeks
  This questionnaire evaluates the quality of sleep
SF12 questionnaire to evaluate the quality of life | At 6 weeks
  This questionnaire evaluates the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No